CLINICAL TRIAL: NCT07063589
Title: Trajectoires Individuelles de Consommation de Cannabis en Situation Habituelle et Observations de Leurs Modalités en Contexte Écologique
Brief Title: Cannabis Use Patterns Among Young Adults and Associations With Social and Health Outcomes.
Acronym: TRICCHOME
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-12297
Record Dates: First submitted 2025-05-12; First posted 2025-07-14 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cannabis Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mobile application — Cannabis use patterns and their resulting subjective experiences, along with social and health-related correlates will be collected in real time using a mobile application specifically designed for this study by a local custom software development company (Osedea, Montreal).

SUMMARY:
The purpose of this study is to identify and characterize patterns of non-therapeutic cannabis consumption and their variation in time in regular/daily users aged 18-24 years using a multi-factor approach (frequency of use, product types, cannabinoid dosages) over a two-year period.

DETAILED DESCRIPTION:
Changes in the legal status of cannabis in Canada have highlighted the need for knowledge about the substance and its effects at individual, population and societal levels. In Quebec, in the past year, one in four cannabis users reported weekly use, and around 15% reported daily use. More specifically, young people between the ages of 18 and 24 account for the largest proportion of this consumption, representing a large proportion of these regular to daily users. Little information is currently available about the correlates, evolution and effects of regular, daily cannabis use in this age group, despite the fact that it is the most widely used in the province.

Such comprehensive longitudinal data on consumption dynamics within this population is crucial for our understanding of whether and how cannabis use trajectories vary over time, characterizing the health and social consequences of cannabis consumption at this critical stage in human development, and ultimately providing evidence for the development of strategies to prevent and mitigate potential harms to this specific population.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 24 years of age;
* Cannabis use frequency of at least 1 day/week in the past three months;
* Ability to speak and read French or English;
* willingness to comply with all study procedures;
* access to a mobile phone.

Exclusion Criteria:

* Planned extended absence during study period (e.g. pending legal action, surgery, incarceration, inpatient residential program) which, in the opinion of the research staff, might prevent completion of the study;
* Current or anticipated treatment for cannabis use disorder, confirmed via self-report;
* Medical document authorizing the use of cannabis for medical purposes;
* Participation in clinical studies or undergoing other investigational procedures involving cannabis or cannabinoids administration.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target population for TRICCHOME is young adults between 18 and 24 years of age, who use cannabis regularly or daily.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Cannabis use patterns | Baseline
  Primary outcome measures of this study are specific assessments of cannabis use patterns, measured at baseline and daily using the mobile app. Primary outcome assessments related to cannabis use patterns will be tracked daily, taking advantage of a short but detailed series of questions taking approximately 1-5 minutes to answer, depending on the number of consumption events during the day. Participants will be advised to provide information even during non-consumption days, which in these cases will be limited to their general appreciation of the day, in addition to the fact that they did not consume that day. Participants will be able to retrospectively enter daily cannabis consumption data up to a maximum of seven days in the past, to minimize recall bias.
Trajectories of consumption patterns over time_Route of administration | From baseline (Day 1) up to two year (Day 730)
  The investigators will use weekly reports on participants' habits surrounding cannabis use in the form of logbook entries, covering the route of administration for each product. This information will be collected for each consumption session during a use day.
Trajectories of consumption patterns over time_product type | From baseline (Day 1) up to two year (Day 730)
  The investigators will use weekly reports on participants' habits surrounding cannabis use in the form of logbook entries, covering the product type for each product. This information will be collected for each consumption session during a use day.
Trajectories of consumption patterns over time_THC constituent (%) | From baseline (Day 1) up to two year (Day 730)
  The investigators will use weekly reports on participants' habits surrounding cannabis use in the form of logbook entries, covering the THC constituent (%) for each product. This information will be collected for each consumption session during a use day.
Trajectories of consumption patterns over time_CBD constituent (%) | From baseline (Day 1) up to two year (Day 730)
  The investigators will use weekly reports on participants' habits surrounding cannabis use in the form of logbook entries, covering the CBD constituent (%) for each product. This information will be collected for each consumption session during a use day.
Trajectories of consumption patterns over time_amount per use | From baseline (Day 1) up to two year (Day 730)
  The investigators will use weekly reports on participants' habits surrounding cannabis use in the form of logbook entries, covering the amount per use for each product. This information will be collected for each consumption session during a use day.
Trajectories of consumption patterns over time_supply source | From baseline (Day 1) up to two year (Day 730)
  The investigators will also capture information on supply source (choices are: cultivated by me or for me, family member or friend or acquaintance, SQDC, legal source from another province, health Canada licensed producer, illegal market) for each product used in the logbook.

SECONDARY OUTCOMES:
Socio-demographic and behavioral determinants | From baseline (Day 1) up to two year (Day 730) and from week 1 to week 104 and every 4 months (Weeks16, 32, 48, 64, 96)
  In addition to the information contained in the weekly logbook entries, for each cannabis use event we will collect socio-demographic variables to identify patterns of cannabis consumption.
  Based on this multi-factor approach, we hypothesize that users will fall into distinct clusters of consumption patterns (e.g., stable, chaotic/variable patterns, etc.), which will each be associated with specific psychosocial determinants and health outcomes.
Socio-demographic and behavioral determinants | At Weeks 16, 32, 48, 64 and 96
  In addition to the information contained in the weekly logbook entries, for each cannabis use event and every four months, various social and health measures will be collected with the mobile application.
  Based on this multi-factor approach, we hypothesize that users will fall into distinct clusters of consumption patterns (e.g., stable, chaotic/variable patterns, etc.), which will each be associated with specific psychosocial determinants and health outcomes.

OTHER OUTCOMES:
Association between variations in cannabis use patterns and health-related and social outcomes. | baseline, Weeks 16, 32, 48, 64 and 96
  The following health-related outcomes will be measured at baseline and at 4-month intervals using the mobile app for a total of nine times.
  Genetic profiles of participant will be used to perform genotype to phenotype associations based on health-related outcomes. Participants will be genotyped at more than 700,000 genome-wide loci to determine if specific genetic variants are significantly associated with some of the patterns of use detected in objective 1. Associations between genetic variants and health-related outcomes will additionally be tested to identify potential genetic vulnerabilities to higher risks of experiencing health problems.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras-Aswad, MD, MS, Principal Investigator — CRCHUM
Locations (1):
- Centre de recherche du Centre Hospitalier Universitaire de Montréal, Montreal, Quebec, Canada